CLINICAL TRIAL: NCT04925531
Title: Antibiotic Use in Facial Fracture Post Injury
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 042.TRA.2016.D
Record Dates: First submitted 2019-08-12; First posted 2021-06-14 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries | interventions — Anti-Bacterial Agents; Ampicillin; Cefazolin; Erythromycin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antibiotic use for <3 days: a retrospective chart review to examine if either the utility of antibiotics administered for 3 days make a difference in the clinical outcomes after facial fractures
  Interventions: Drug: Antibiotics
- Antibiotic use for 5 days: a retrospective chart review to examine if either the utility of antibiotics administered for 5 days make a difference in the clinical outcomes after facial fractures
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — to examine if either the utility of antibiotics administered for 3 days or 5 days make a difference in the clinical outcomes after facial fractures in trauma patients.
  Other Names: Ampicillin, Ancef, Erythro

SUMMARY:
Facial fractures make up a significant proportion of injuries in trauma patients (1, 2). Approximately 3 million individuals suffer craniofacial trauma in the United States on a yearly basis, and approximately 50% of all wounds presenting to emergency rooms involve the head and neck (1, 2). Treatment of these fractures often results in standard surgical interventions. While up to the early 1980's perioperative antibiotic prophylaxis in maxillofacial surgery was controversial, its efficacy is well accepted today (3). Previous research work showed that the administration of antibiotics one hour preoperatively and eight hours after the intervention reduces the incidence of infectious complications in facial fractures from 42.2% to 8.9% (4). However there is still no consensus about the duration of the postoperative administration. In literature postoperative prophylaxis in facial fractures varies from single-shot up to duration of 7 and even ten days postoperatively. The use of antibiotics can be associated with allergic or toxic reactions, adverse effects, drug interactions and increasing bacterial resistance (5). In addition some authors assume that a prolonged administration of antibiotics might increase the risk of infectious complications via superinfection. On the other hand a short term or single shot administration might not be enough to prevent the onset of a postoperative infection. Up to date there is no standard to support the duration of antibiotic administration after surgical repair of a facial fracture. In this proposal, Investigators are aiming to investigate if either the utility of antibiotics administered for 3 days or 5 days make a difference in the clinical outcomes after facial fractures.

DETAILED DESCRIPTION:
This proposed research is a retrospective chart review to examine if either the utility of antibiotics administered for 3 days or 5 days make a difference in the clinical outcomes after facial fractures.

Records of trauma patients who were admitted to Methodist Health System (MHS) between January1st 2010 and December 31st 2015 will be retrieved to review the clinical charts according to our inclusion and exclusion criteria.

Patients will be segregated in to two groups according to the duration of antibiotic use, group 1 (less than 3days) and group 2 (5 days).

Basic demographics and clinical outcomes parameters as noted above will be attained from the patient's medical records.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patient's ≥ 18 years of age.
* Blunt and penetration injury.

Exclusion Criteria:

* Pregnant and breast feeding women.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: trauma patients who were admitted to MHS between January1st 2010 and December 31st 2015
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-07-29; Primary Completion 2024-07-23 (Estimated); Study Completion 2024-07-23 (Estimated)

PRIMARY OUTCOMES:
Injury associated infectious complications within 30-days of injury | 3 days post trauma
  This will help to determine if specific intervals of prophylactic antibiotic use for facial fracture patients decreases the incidence of fracture-associated infections.

SECONDARY OUTCOMES:
Demographics | through study completion, an average of 2 years
  Age, sex, ethnicity

CONTACTS AND LOCATIONS:
Overall Officials: Michael Truitt, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided